CLINICAL TRIAL: NCT03494842
Title: A Doubled Blinded Randomised Controlled Trial of Conscious Sedation With Transcutaneous Nerve Stimulation for Pain Relief During Suction Evacuation for Termination of First Trimester Pregnancies
Brief Title: TENS for Suction Evacuation for Termination of 1st Trimester Pregnancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, KEEDON WONG, Principal Investigator (Dr.), Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW18-008
Record Dates: First submitted 2018-03-05; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Pregnancy, Abdominal; Termination of Pregnancy; Pain, Nerve
Keywords: TENS; pain relief; STOP; surgical abortion
MeSH Terms: conditions — Pregnancy, Abdominal; Neuralgia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After the written informed consent is obtained, subjects will be randomly allocated into one of the two groups: (a) the active TENS group and (b) the placebo TENS group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the active TENS group (Active Comparator): Transcutaneous nerve stimulation (TENS)
  Interventions: Device: Transcutaneous nerve stimulation (TENS)
- the placebo TENS group (Placebo Comparator): Placebo Transcutaneous nerve stimulation (TENS)
  Interventions: Device: Placebo Transcutaneous nerve stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous nerve stimulation (TENS) — The active TENS unit (delivers electrical stimulation) with indicator light
  Other Names: the active TENS group
  Arms: the active TENS group
Device: Placebo Transcutaneous nerve stimulation (TENS) — the placebo TENS unit (delivers no electrical stimulation) with indicator light
  Other Names: the placebo TENS group
  Arms: the placebo TENS group

SUMMARY:
To study the effectiveness of the pain relief method of transcutaneous electrical nerve stimulation (TENS) for women who will undergo suction evacuation under conscious sedation for first trimester termination of pregnancy.

DETAILED DESCRIPTION:
Suction evacuation is a minor gynecological procedure commonly performed at an outpatient setting for termination of pregnancy. Although it is a simple surgical procedure lasting 5-10 min and can be done under various methods of pain control, 78-97% of women still report at least moderate procedural pain, especially during injection of paracervical block, cervical dilation, suction aspiration and postoperatively with uterine cramping. In addition, those pharmacological analgesic methods are often associated with numerous adverse effects and cannot be applicable to all women.

The transcutaneous nerve stimulation (TENS) method is commonly used to treat labour pain. It is an inexpensive, quick, easy to use and noninvasive pain relief method. A recent study by Lison et al. on TENS for office hysteroscopy demonstrated a significant decrease in pain scores when compared to control and placebo groups.

The rationale of TENS lies in achieving pain reduction when electric stimulation alters the nociceptive transmission in the dorsal horn of the spinal cord; this means the electrode has to be adequately applied in the right receptive field of the body to achieve pain control. For the setting of TENS there is evidence supporting superior pain relief by random high frequencies TENS over fixed frequency. Increasing the pulse duration to above 250 microseconds also produces better analgesics effect.

In suction evacuation, the nerve roots of T10-L1 and S2-S4 becomes relevant as they correspond to the nerve supply to the whole uterus and cervix. Lison et al placed electrodes at these levels parallel to the spinal cord in their study and have instructed their subjects to increase the TENS intensity to the maximum nonpainful level, allowing further increase when their stimulus perception decrease as a result of nerve accommodation.

Its use in suction evacuation however, remains undetermined as there is no published study in this area.

ELIGIBILITY:
Inclusion Criteria:

* Chinese aged 18 years or above and mentally competent
* Up to 12 weeks gestation on the day of STOP
* Size of the uterus on pelvic examination compatible with estimated duration of pregnancy, or dating confirmed with ultrasound scan
* Normal general and gynecological examination

Exclusion Criteria:

* Skin damage or allergy at site of TENS pads application
* Previous experience with TENS
* History of pacemarker insertion
* History of severe respiratory or cardiac disease
* Severe and recurrent liver disease
* Allergic to lignocaine
* Myasthenia gravis
* Psychiatric conditions requiring medication
* Disorders that constitute contraindications to use of prostaglandins

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who has up to 12 weeks gestation on the day of STOP
Enrollment: 170 (Estimated)
Dates: Start 2018-04-26 (Estimated); Primary Completion 2020-01-22 (Estimated); Study Completion 2020-03-22 (Estimated)

PRIMARY OUTCOMES:
To assess the change of 100-point visual analogue pain scale in 3 time points | Patient will be asked for the pain intensity by using the 100 mm linear VAS 5 minutes before receiving the active TENS/ placebo TENS before the start of suction evacuation, reassess 20 minutes later and 1 hour after operation.
  To measure patient's pain intensity before and after suction TOP by using The Visual Analogue Scale (VAS) consists of a straight line length of 100 mm with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain. This tool was first used in psychology by Freyd in 1923.

SECONDARY OUTCOMES:
To assess the change of Anxiety level of the patients in 3 time points by using State-Trait Anxiety Inventory Questionnaire to record patient's anxiety level. | Patient will be asked for the anxiety level by using STAI 5 minutes before receiving the active TENS/ placebo TENS before the start of suction evacuation, reassess 20 minutes later and 1 hour after operation.
  To record patient's anxiety level for comparison
To assess the difficulty of the operation | The surgeon will be asked to fill the assessment form right after the suction evacuation operation immediately.
  The surgeon will assess the difficulty of the operation by using LEVEL OF SEDATION AND DIFFICULTY OF OPERATION ASSESSMENT FORM (proposed by Ramsay et al.)

CONTACTS AND LOCATIONS:
Overall Officials: Keedon Wong, MBBS, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Belanger E, Melzack R, Lauzon P. Pain of first-trimester abortion: a study of psychosocial and medical predictors. Pain. 1989 Mar;36(3):339-350. doi: 10.1016/0304-3959(89)90094-8. PMID 2710563
- [Background] Wong CY, Ng EH, Ngai SW, Ho PC. A randomized, double blind, placebo-controlled study to investigate the use of conscious sedation in conjunction with paracervical block for reducing pain in termination of first trimester pregnancy by suction evacuation. Hum Reprod. 2002 May;17(5):1222-5. doi: 10.1093/humrep/17.5.1222. PMID 11980742
- [Background] Lison JF, Amer-Cuenca JJ, Piquer-Marti S, Benavent-Caballer V, Bivia-Roig G, Marin-Buck A. Transcutaneous Nerve Stimulation for Pain Relief During Office Hysteroscopy: A Randomized Controlled Trial. Obstet Gynecol. 2017 Feb;129(2):363-370. doi: 10.1097/AOG.0000000000001842. PMID 28079781
- [Background] Vance CG, Dailey DL, Rakel BA, Sluka KA. Using TENS for pain control: the state of the evidence. Pain Manag. 2014 May;4(3):197-209. doi: 10.2217/pmt.14.13. PMID 24953072
- [Background] Sluka KA, Walsh D. Transcutaneous electrical nerve stimulation: basic science mechanisms and clinical effectiveness. J Pain. 2003 Apr;4(3):109-21. doi: 10.1054/jpai.2003.434. PMID 14622708